CLINICAL TRIAL: NCT04395508
Title: An Expanded Access, Single-Arm, Multicenter Study to Provide at Home Subcutaneous Administration of Pertuzumab and Trastuzumab Fixed-Dose Combination (PH FDC SC) for Patients With HER2-Positive Breast Cancer During the COVID-19 Pandemic
Brief Title: An Expanded Access Study to Provide at Home Subcutaneous Administration of Pertuzumab and Trastuzumab Fixed-Dose Combination (PH FDC SC) for Patients With HER2-Positive Breast Cancer During the COVID-19 Pandemic
Status: Approved for marketing | Type: Expanded Access
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AL42478
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pertuzumab; Trastuzumab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Pertuzumab and Trastuzumab Fixed-Dose Combination for Subcutaneous Administration (PH FDC SC) — PH FDC SC is given as a fixed dose (i.e. non-weight based) subcutaneous injection. Two dosage configurations of PH FDC SC may be administered in the study: a 15-millilitre (mL) loading dose consisting of 1200 milligrams (mg) pertuzumab and 600 mg trastuzumab and a 10-mL maintenance dose consisting of 600 mg pertuzumab and 600 mg trastuzumab. Participants who have had ≥6 weeks since their last P+H IV, PH FDC SC, or are receiving trastuzumab SC treatment must receive a loading dose before continuing with maintenance doses for subsequent administrations. Note that participants receiving trastuzumab SC only (i.e. without pertuzumab) must receive a loading dose regardless of time since last treatment.
  Other Names: Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf; PHESGO®; RO7198574; RG6264

SUMMARY:
This single arm, multicenter study provides the pertuzumab and trastuzumab fixed-dose combination formulation for subcutaneous injection (PH FDC SC) administered at home by a home health nursing provider for patients with human epidermal growth factor receptor 2-positive (HER2+) breast cancer who have completed concurrent chemotherapy with pertuzumab (Perjeta) and trastuzumab (Herceptin) by intravenous administration (P+H IV) and are currently receiving or will be receiving maintenance therapy with P+H IV, PH FDC SC, or trastuzumab SC in the clinic. The main objective is to enable continuity of care during the COVID-19 pandemic.

This study will enroll approximately 200 patients in the United States.

Participants with early or metastatic HER2+ breast cancer will be enrolled in this study. Participants with metastatic HER2+ breast cancer will receive treatment every 3 weeks and continue treatment unless early cessation is necessary due to disease recurrence, disease progression, unacceptable toxicity, participant withdrawal of consent, or per physician's recommendation. Participants with early HER2+ breast cancer will receive PH FDC SC to complete 1 year (up to 18 cycles) of dual blockade, including the P+H IV, PH FDC SC, or trastuzumab SC they received prior to enrolling in this study, unless early cessation is necessary due to disease recurrence, disease progression, unacceptable toxicity, participant withdrawal of consent, or per physician's recommendation.

A remote cardiac surveillance substudy will be optional for patients enrolled at select sites.

The Sponsor may decide to terminate the study when the COVID-19 pandemic is no longer a risk for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients with histologically confirmed human epidermal growth factor receptor 2-positive (HER2+) breast cancer who have completed chemotherapy in combination with P+H IV and are currently receiving or will be receiving maintenance P+H IV, PH FDC SC, or trastuzumab SC (regardless of remaining treatment cycles [e.g., only 1 cycle remaining])
* HER2+ status must have been previously determined and is defined as 3+ by immunohistochemistry (IHC) and/or positive by HER2 amplification by in situ hybridization (ISH) with a ratio of ≥2 for the number of HER2 gene copies to the number of chromosome 17 copies
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Intact skin at planned site of subcutaneous (SC) injections (thigh)
* Baseline and most recent (within 3 months) LVEF ≥ 50% measured by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA)
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating eggs, as defined in the protocol
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined in the protocol

Exclusion Criteria:

* Current or prior history of active malignancy (other than current breast cancer) within the last 5 years. Appropriately treated non-melanoma skin cancer; in situ carcinomas, including cervix, colon, or skin; or Stage I uterine cancer within the last 5 years are allowed
* Investigational treatment within 4 weeks of enrollment
* Patients with any severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infections should not be enrolled in the trial (in the current situation, this also applies to patients with suspected or confirmed COVID-19 infection). Patients with suspected or confirmed COVID-19 may be re-screened for eligibility following physician-prescribed COVID-19 treatment and/or a quarantine period consistent with current Centers for Disease Control and Prevention (CDC) guidelines.
* Patients who may have had a recent episode of thromboembolism and are still trying to optimize the anticoagulation dose and/or have not normalized their INR
* Serious cardiac illness or medical conditions
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias, such as structural heart disease (e.g., severe left ventricular systolic dysfunction [LVSD], left ventricular hypertrophy), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or long QT syndrome
* Inadequate bone marrow function
* Impaired liver function
* Renal function with creatinine clearance <50 mL/min using the Cockroft-Gault formula
* Major surgical procedure unrelated to breast cancer within 28 days prior to study entry or anticipation of the need for major surgery during the course of study treatment
* Current severe, uncontrolled systemic disease that may interfere with planned treatment (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease; wound-healing disorders)
* Pregnant or breastfeeding, or intending to become pregnant during the study or within seven months after the last dose of study treatment
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in, and completion of, the study
* Known active liver disease, for example, active viral hepatitis infection (i.e., hepatitis B or hepatitis C), autoimmune hepatic disorders, or sclerosing cholangitis
* Concurrent, serious, uncontrolled infections, or known infection with human immunodeficiency virus (HIV)
* Known hypersensitivity to any of the study drugs, excipients, and/or murine proteins or a history of severe allergic or immunological reactions, e.g. difficult to control asthma
* Previously experienced severe injection related reactions with P+H IV, PH FDC SC, and/or trastuzumab SC
* Current chronic daily treatment with corticosteroids (dose >10 mg methylprednisolone or equivalent excluding inhaled steroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (12):
- United States (12):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - UCSF Helen Diller Family CCC, San Francisco, California
  - Stanford Univ School of Med; Oncology, Stanford, California
  - University Of Colorado, Aurora, Colorado
  - MedStar Washington Hosp Center, Washington D.C., District of Columbia
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Hospital-Rochester, St. Marys Campus - PPDS, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington